CLINICAL TRIAL: NCT04521413
Title: A First-In-Human, Phase 1/2 Study Of CFI-402411, a Hematopoietic Progenitor Kinase-1 (HPK1) Inhibitor, as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Malignancies
Brief Title: Safety and Efficacy Study of CFI-402411 in Subjects With Advanced Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treadwell Therapeutics, Inc (Industry)
Collaborators: TIO Discovery Engine (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWT-101
Record Dates: First submitted 2020-07-31; First posted 2020-08-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Malignancies
Keywords: advanced tumors; pembro; keytruda; pembrolizumab; 2411; CFI-402411; first in human; first-in-human; hematopoietic progenitor kinase-1 inhibitor; HPK1; advanced solid malignancies; solid malignancies; TWT-101; TWT101; UHN; University Health Network; Treadwell Therapeutics
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion for monotherapy and combination arms with pembrolizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A1: Monotherapy Escalation (Experimental): Dose escalation arm with CFI-402411. CFI-402411 is administered orally once daily.
  Interventions: Drug: CFI-402411
- A2: Monotherapy Biomarker (Experimental): Dose escalation biomarker arm with CFI-402411. CFI-402411 is administered orally once daily.
  Interventions: Drug: CFI-402411
- A3: Monotherapy Expansion (Experimental): Dose expansion arm with CFI-402411 at its recommended phase 2 dose.
  Interventions: Drug: CFI-402411
- B1: Combination Escalation (Experimental): Dose escalation arm with CFI-402411 in combination with pembrolizumab (at its labeled dose and schedule).
  Interventions: Drug: CFI-402411; Drug: Pembrolizumab
- B2: Combination Expansion (Experimental): Dose expansion arm with the recommended phase 2 dose of CFI-402411 in combination with pembrolizumab (at its labeled dose and schedule).
  Interventions: Drug: CFI-402411; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CFI-402411 — CFI-402411 is administered orally once daily. The starting dose is 80 mg/day for escalation arms and the recommended dose for the expansion arms.
  Other Names: 2411; 402411
Drug: Pembrolizumab — Pembrolizumab will be given at its labeled dose and schedule, 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks.
  Other Names: Keytruda; pembro
  Arms: B1: Combination Escalation; B2: Combination Expansion

SUMMARY:
The purpose of this study is to test the safety of an investigational drug called CFI-402411 alone and in combination with pembrolizumab and to study its effects in patients with advanced solid tumors who have progressed following previous therapies.

DETAILED DESCRIPTION:
This study will be a first-in-human study evaluating the safety and tolerability of CFI-402411 in subjects with advanced solid malignancies, when CFI-402411 is administered as a single agent or in combination with pembrolizumab. CFI-402411 is an oral pill that blocks the function of HPK1. Blocking HPK1 could stimulate an immune response against the tumor in patients. This immune response could be further enhanced when combined with pembrolizumab. The data obtained from this study will determine the dose and schedule and subject selection for further clinical studies.

Pre-clinical findings support further development of CFI-402411 as a novel anti-cancer agent, and the combination of CFI-402411 with pembrolizumab as a potential strategy to improve outcomes of subjects with advanced malignancies.

ELIGIBILITY:
Key Inclusion Criteria: Study-Wide Eligibility (Across All Study Parts):

1. Age > 18 years old
2. Have progressed after ≥ 1, but no more than 3 regimens of systemic therapies for recurrent / metastatic disease.
3. Subjects must have measurable disease.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Part A1: Monotherapy Dose Escalation Inclusion Criteria

1. Histological or cytological confirmation of advanced solid malignancy that is refractory to or not a candidate for current standard treatment(s) and for whom no standard therapy is available.

Part A2: Biomarker-Focused Monotherapy Backfills Inclusion Criteria

1. Histological or cytological confirmation of one of the advanced cancers listed below;

   * NSCLC
   * SCLC
   * cutaneous melanoma
   * Merkel cell carcinoma
   * squamous cell carcinoma of head and neck, anal canal, or skin
   * urothelial cancer
   * clear cell or non-clear cell renal cell carcinoma
   * triple negative breast cancer
   * endometrial cancer (regardless of MSI status)
   * cervical cancer
   * gastroesophageal cancer
   * hepatocellular cancer
   * any histology if known to be microsatellite-instability high (MSI-H)
2. Tumors must be refractory to or not a candidate for current standard treatment(s) and for whom no standard therapy exists.

Part A3: Monotherapy Expansion Inclusion Criteria

1. Histological or cytological confirmation of one of the advanced cancers listed below;

   * NSCLC cancer any histology
   * SCLC
   * cutaneous melanoma
   * Merkel cell carcinoma
   * squamous cell carcinoma of head and neck, anal canal, or skin
   * urothelial cancer
   * clear cell or non-clear cell renal cell carcinoma
   * triple negative breast cancer
   * endometrial cancer (regardless of MSI status)
   * cervical cancer
   * gastroesophageal cancer
   * hepatocellular
   * any histology if known to be microsatellite-instability high (MSI-H)
2. Tumors must be refractory to or subjects intolerant of current standard treatment(s) and for whom no standard therapies are available.
3. Optional biopsies: Subjects that consent to optional fresh tumor biopsies must have at least one non-target soft tissue tumor lesion that can be biopsied.

Part B1: CFI-402411 in Combination with Pembrolizumab Dose Escalation Inclusion Criteria

1. Subjects must be deemed eligible by the Investigator to receive pembrolizumab.
2. Histological or cytological confirmation of one of the advanced cancers listed below (list may vary in each country, USA shown here);

   * NSCLC cancer any histology
   * SCLC
   * cutaneous melanoma
   * Merkel cell carcinoma
   * squamous cell carcinoma of head and neck, anal canal, or skin
   * urothelial cancer
   * clear cell or non-clear cell renal cell carcinoma
   * triple negative breast cancer
   * endometrial cancer (regardless of MSI status)
   * cervical cancer
   * gastroesophageal cancer
   * hepatocellular cancer
   * any histology if known to be microsatellite-instability high (MSI-H)

Tumors must be refractory to or subjects intolerant of current standard treatment(s) or for whom no standard therapy is available.

Part B2: CFI-402411 in Combination with Pembrolizumab Expansion Inclusion Criteria

1. Subjects must be deemed eligible by the Investigator to receive pembrolizumab
2. Histological or cytological confirmation of one of the advanced cancers listed below (list may vary in each country, USA shown here);

   * non-small cell lung cancer any histology
   * SCLC
   * cutaneous melanoma
   * Merkel Cell carcinoma
   * squamous cell carcinoma of head and neck, anal canal, or skin
   * urothelial cancer
   * clear cell or non-clear cell renal cell carcinoma
   * triple negative breast cancer
   * endometrial cancer (regardless of MSI status)
   * gastroesophageal cancer
   * hepatocellular cancer
   * any histology if known to be microsatellite-instability high (MSI-H)
3. Tumors must be refractory to or subjects intolerant of current standard non-IO treatment(s) or for whom no standard therapy is available.

Key Exclusion Criteria: Study-Wide Eligibility (Across All Study Parts)

Subjects will be excluded from the study if any of the following criteria is met;

1. Previous treatment with an HPK1 inhibitor in other clinical trials.
2. Diagnosis of autoimmune-based disease or clinically significant auto-immune disorders.
3. Have symptomatic congestive heart failure, active angina pectoris or recent myocardial infarction (within 6 mos).
4. Have chronic atrial fibrillation.
5. Known central nervous system metastasis.
6. Stroke or transient ischemic attack, or other ischemic events or thromboembolic events within 3 months of study enrollment.
7. A history of QTc prolongation or a marked baseline prolongation of QT/QTc interval or a history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of adverse events of CFI-402411 as a single agent and at the recommended phase 2 dose (RP2D). | 48 months
  The number of subjects who experience an adverse event that was possibly related to study drug.
To assess the incidence of adverse events with CFI-402411 in combination with pembrolizumab and at the RP2D. | 48 months
  The number of subjects who experience an adverse event that was possibly related to study drug.
To examine best overall response rate in subjects treated at multiple dose levels of CFI-402411. | 48 months
  Best overall response rate will be summarized by dose cohort and overall using the percent of patients in each tumor response category.
To examine progression free survival in subjects treated at multiple dose levels of CFI-402411. | 48 months
  Time from first dose to disease progression or death whichever occurs first will be calculated and summarized for all patients by dose cohort and overall.

SECONDARY OUTCOMES:
To identify the maximum tolerated dose of single agent CFI-402411 alone and in combination with pembrolizumab. | 48 months
  Safety tables and pharmacokinetic tables will be assessed.
To further assess the incidence of adverse events of CFI-402411. | 48 months
  The number of subjects who experience an adverse event that was possibly related to study drug.
To assess best overall response of CFI-402411 monotherapy and in combination with pembrolizumab. | 48 months
  Best overall response rate will be summarized by dose cohort and overall using the percent of patients in each tumor response category.
To assess overall response rates of CFI-402411 monotherapy and in combination with pembrolizumab. | 48 months
  For all subjects the overall response rates of complete response and partial response will be calculated and summarized by dose cohort and overall.
To assess overall survival of CFI-402411 monotherapy and in combination with pembrolizumab. | 48 months
  The time from first dose until the date of death from any cause will be calculated and summarized for all patients by dose cohort and overall.
To assess progression free survival of CFI-402411 monotherapy and in combination with pembrolizumab. | 48 months
  Time from first dose to disease progression or death whichever occurs first will be calculated and summarized for all patients by dose cohort and overall.
To assess duration of response of CFI-402411 monotherapy and in combination with pembrolizumab. | 48 months
  The time from the first objective response to the time of documented disease progression or death due to any cause, whichever occurs first, will be calculated and summarized for all patients by dose cohort and overall.
To assess the pharmacokinetic profile of CFI-402411 alone when it is administered in combination with pembrolizumab through AUC. | 48 months
  Area under the plasma concentration (AUC) versus time curve from time 0 to time of least measurable concentration tabulated by dose group.
To assess the pharmacokinetic profile of CFI-402411 alone when it is administered in combination with pembrolizumab through Cmax. | 48 months
  Cmax will be assessed through the maximum measured plasma concentration occurring at Tmax tabulated by dose group.
To assess the pharmacokinetic profile of CFI-402411 alone when it is administered in combination with pembrolizumab through Tmax. | 48 months
  Tmax will be assessed by the time to achieve maximum plasma concentration and will be tabulated by dose group.
To assess the pharmacokinetic profile of CFI-402411 alone when it is administered in combination with pembrolizumab though Cmin. | 48 months
  Cmin will be calculated through the measured pre-dose plasma concentration and tabulated by dose group.
To assess the pharmacokinetic profile of CFI-402411 alone when it is administered in combination with pembrolizumab through T1/2. | 48 months
  Elimination half life will be calculated and tabulated by dose group.
To evaluate the effect of CFI-402411 treatment on immune- or disease related biomarkers. | 48 months
  The effects of CFI-402411 on pharmacodynamic biomarkers (cytokine levels) will be assessed by percent changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Omid Hamid, Dr, Principal Investigator — The Angeles Clinic, Los Angeles
Locations (13):
- United States (9):
  - University of California San Diego, La Jolla, California
  - The Angeles Clinic, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Sarasota, Florida
  - START - Mid-West, Grand Rapids, Michigan
  - SCRI - Nashville, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - START - San Antonio, San Antonio, Texas
  - Virginia Cancer Specialist, Fairfax, Virginia
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It is too early to determine whether we will make IPD available - we do not yet have a process written on this. Field will be updated once our policy / process is written.